CLINICAL TRIAL: NCT05950412
Title: Relationship Between Pitch Discrimination, Music Abilities and Emotional Speech Perception in School Aged Children With Cochlear Implant
Brief Title: Paraverbal Components of Language and Cochlear Implant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5427
Record Dates: First submitted 2023-07-10; First posted 2023-07-18 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-06

CONDITIONS: Hearing Loss, Sensorineural
Keywords: Paraverbal Components of Language and Cochlear Implant
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators evaluated patients older than 6 years old, with severe hearing loss, cochlear implant wearers, able to perform a series of tests (TUISE, the pitch discrimination test, the melody discrimination test, VAS) to assess the skills of perceiving spectral components of music and understanding emotional states of language investigating the relationship between musical ability, pitch discrimination and paraverbal language comprehension.

DETAILED DESCRIPTION:
The investigators evaluated patients with severe hearing loss, undergoing cochlear impantation, to assess the skills of perceiving spectral components of music and understanding emotional states of language.

Each patient will undergo:

1. Music test: a battery of music tests has been designed to assess CI-mediated music perception. The software will be installed on a computer, which is normally used to adapt patients' maps in routine adaptation sessions. It consists of two parts: A) the pitch discrimination test; B) the melody discrimination test

   A) In the pitch discrimination test, the stimuli consist of pairs of notes played by a piano and spaced at least one semitone apart, semitone being the smallest interval in traditional Western music. The notes are distributed within the middle three octaves (C4, C5, C6, each corresponding to the following frequency bands: 262 Hz-523 Hz, 523 Hz-1046 Hz, and 1046 Hz- 1976 Hz), used for most of the pieces, for a total of 36 notes. After listening to each pair of notes, the patient is asked to indicate whether they are the same or different in pitch. It consists of seven levels of increasing difficulty determined by the reduction in the distance between notes: the 1st level included pairs of notes 12 semitones apart (easiest task), while the 7th level included notes one semitone apart (most difficult task). Each level is further divided into two tests: TEST A: consisting of two parts (each of 10 questions) in which the subject must choose between 2 notes belonging to the 5th and 6th musical octaves (523-1976 Hz). TEST B: consists of two parts (each of 10 questions) in which the subject must choose between 2 notes belonging to the 4th and 5th musical octaves (262-988 Hz). In the last 2 levels (6th and 7th levels) there are 20 more questions investigating discrimination on the middle (related to the 5th octave). At the end the score of each level will be calculated (as the percentage of correct answers) and the final total score.

   B) The melody discrimination test consists of 6 popular cartoon songs in digital recording, synthesized with Finale™ 2008 (MakeMusic Inc., Eden Prairie, MN). Before the test performance, subjects will be asked to watch a 30-second cartoon scene and memorize the corresponding song from an IBM© laptop (IBM, Armonk, USA). Each song will be presented twice, for a total of 12 entries. The music test is divided into two sessions: in session 1, full version songs (instrumental plus vocal) for a total of 6 voices. Patients will indicate the distinctive character on the screen for each song. In session 2, songs in melodic version, presented in random order for a total of 6 musical items. An overall score will be calculated based on the correctly identified elements.
2. TUISE test (Auditory Test Identifying Emotional States): the Auditory Test of Identifying Emotional States (T.U.I.S.E.) is a new instrument to assess emotional states. It consists of 4 subtests, each consisting of 15 questions. Each item involves an audio recording of short sentences spoken with varying intonation by different readers of both sexes. To ensure proper administration, all background noise was removed and semantically neutral sentences were chosen. In addition, a glossary was developed with explanations and examples for all the emotional states presented. In the 1st subtest, the task is to identify among the four basic emotions (happy, sad, angry, scared) which one best described the speaker's emotional state (only one term, among the four words, correctly represented what the speaker was thinking or feeling). In the 2nd subtest, more complex emotions are assessed as patients have to identify among four terms regarding complex emotional states varied for each item, the one that correctly expressed the emotional state expressed by the speaker (joking, doubtful, agitated, rude, concerned, friendly, bored, excited, hopeful, surprised, overbearing and angry). In the 3rd subtest, which required speaker discrimination, each item consisted of two recordings. They are, in fact, presented with several pairs of vocal traces, and the patient has to distinguish whether each item is presented by different people or not. Finally, the 4th subtest consists to identify the gender of the speaker. Each item consists of an audio track and the patient have to mark whether the speaker is male or female.
3. Visual analog scale (VAS scale): it is used to estimate, with a score from 1 to 10, how pleasant it is to listen to music.

The aim is to investigate the relationship between musical ability, pitch discrimination and paraverbal language comprehension.

ELIGIBILITY:
Inclusion Criteria:

* patients with severe-profound sensorineural hearing loss undergoing cochlear implantation at Fondazione Policlinico Universitario A. Gemelli-IRCCS, Rome, Italy;
* Intracochlear implant placement in soft surgery technique, by mastoidectomy and posterior tympanotomy and insertion of the electrode array through the round window
* age >6 years
* patients without associated disabilities, with good auditory verbal perceptual skills and adequate language skills
* the ability to understand and perform the tests administered

Exclusion Criteria:

* pulsating tinnitus
* congenital malformation of the auditory system
* history of vestibular schwannoma, active middle ear disease and complete ossification of the cochlea.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing cochlear implantation, able to understand and perform the test administered.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Pitch discrimination test | 6 months after cochlear implantation
  The stimuli consist of pairs of notes played by a piano and spaced at least one semitone apart, semitone being the smallest interval in traditional Western music. The patient is asked to indicate whether they are the same or different in pitch. It assesses discriminative skills
Melody discrimination test | 6 months after cochlear implantation
  Consists of 6 popular cartoon songs in digital recording. Subjects will be asked to watch a 30-second cartoon scene and memorize the corresponding song. In session 1, full version songs (instrumental plus vocal) for a total of 6 voices. Patients will indicate the distinctive character on the screen for each song. In session 2, songs in melodic version, presented in random order for a total of 6 musical items. It assesses discriminative skills
TUISE (Auditory Test of Identifying Emotional States) | 6 months after cochlear implantation
  is a new instrument to assess emotional states. It consists of 4 subtests, each consisting of 15 questions. Each item involves an audio recording of short sentences spoken with varying intonation by different readers of both sexes. To ensure proper administration, all background noise was removed and semantically neutral sentences were chosen. In addition, a glossary was developed with explanations and examples for all the emotional states presented.
VAS | 6 months after cochlear implantation
  to estimate, with a score from 1 to 10, how pleasant it is to listen to music

CONTACTS AND LOCATIONS:
Overall Officials: Walter Di Nardo, Professor, Principal Investigator — Fondazione Universitaria Policlinico Agostino Gemelli IRCCS
Locations (1):
- Fondazione Universitaria Policlinico Agostino Gemelli IRCCS, Rome, Lazio, Italy

REFERENCES:
- [Result] Issing C, Baumann U, Pantel J, Stover T. Cochlear Implant Therapy Improves the Quality of Life in Older Patients-A Prospective Evaluation Study. Otol Neurotol. 2020 Oct;41(9):1214-1221. doi: 10.1097/MAO.0000000000002741. PMID 32925841
- [Result] Di Nardo W, Anzivino R, Giannantonio S, Schinaia L, Paludetti G. The effects of cochlear implantation on quality of life in the elderly. Eur Arch Otorhinolaryngol. 2014 Jan;271(1):65-73. doi: 10.1007/s00405-013-2396-1. Epub 2013 Feb 15. PMID 23411946
- [Result] Qazi OU, van Dijk B, Moonen M, Wouters J. Understanding the effect of noise on electrical stimulation sequences in cochlear implants and its impact on speech intelligibility. Hear Res. 2013 May;299:79-87. doi: 10.1016/j.heares.2013.01.018. Epub 2013 Feb 8. PMID 23396271
- [Result] Kressner AA, May T, Dau T. Effect of Noise Reduction Gain Errors on Simulated Cochlear Implant Speech Intelligibility. Trends Hear. 2019 Jan-Dec;23:2331216519825930. doi: 10.1177/2331216519825930. PMID 30755108
- [Result] Jiam NT, Caldwell MT, Limb CJ. What Does Music Sound Like for a Cochlear Implant User? Otol Neurotol. 2017 Sep;38(8):e240-e247. doi: 10.1097/MAO.0000000000001448. PMID 28806333
- [Result] Jiam NT, Limb CJ. Rhythm processing in cochlear implant-mediated music perception. Ann N Y Acad Sci. 2019 Oct;1453(1):22-28. doi: 10.1111/nyas.14130. Epub 2019 Jun 6. PMID 31168793
- [Result] Nardo WD, Cantore I, Cianfrone F, Melillo P, Fetoni AR, Paludetti G. Differences between electrode-assigned frequencies and cochlear implant recipient pitch perception. Acta Otolaryngol. 2007 Apr;127(4):370-7. doi: 10.1080/00016480601158765. PMID 17453456
- [Result] Vermeire K, Landsberger DM, Van de Heyning PH, Voormolen M, Kleine Punte A, Schatzer R, Zierhofer C. Frequency-place map for electrical stimulation in cochlear implants: Change over time. Hear Res. 2015 Aug;326:8-14. doi: 10.1016/j.heares.2015.03.011. Epub 2015 Apr 1. PMID 25840373
- [Result] Canfarotta MW, Dillon MT, Buss E, Pillsbury HC, Brown KD, O'Connell BP. Frequency-to-Place Mismatch: Characterizing Variability and the Influence on Speech Perception Outcomes in Cochlear Implant Recipients. Ear Hear. 2020 Sep/Oct;41(5):1349-1361. doi: 10.1097/AUD.0000000000000864. PMID 32205726
- [Result] Di Nardo W, Scorpecci A, Giannantonio S, Cianfrone F, Parrilla C, Paludetti G. Cochlear implant patients' speech understanding in background noise: effect of mismatch between electrode assigned frequencies and perceived pitch. J Laryngol Otol. 2010 Aug;124(8):828-34. doi: 10.1017/S0022215110000320. Epub 2010 Mar 5. PMID 20202276
- [Result] Di Nardo W, Scorpecci A, Giannantonio S, Cianfrone F, Paludetti G. Improving melody recognition in cochlear implant recipients through individualized frequency map fitting. Eur Arch Otorhinolaryngol. 2011 Jan;268(1):27-39. doi: 10.1007/s00405-010-1335-7. Epub 2010 Jul 16. PMID 20635091
- [Result] Di Nardo W, Schinaia L, Anzivino R, De Corso E, Ciacciarelli A, Paludetti G. Musical training software for children with cochlear implants. Acta Otorhinolaryngol Ital. 2015 Oct;35(4):249-57. PMID 26824211